CLINICAL TRIAL: NCT06799416
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of ARGX-109 Administered Subcutaneously in Healthy Adult Participants
Brief Title: A Study to Assess the Safety of ARGX-109 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARGX-109-2401
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARGX-109 (Experimental): Participants receiving the experimental drug
  Interventions: Biological: ARGX-109
- Placebo (Placebo Comparator): Participants receiving placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARGX-109 — administrations of ARGX-109
  Arms: ARGX-109
Other: Placebo — administrations of placebo comparator
  Arms: Placebo

SUMMARY:
This study aims to assess the safety of ARGX-109 in healthy adults. Another aim is to measure the amount of ARGX-109 in the blood over time to learn how it moves through the body and acts in the body. Each participant will remain in the study for approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* is aged 18 to 65 years, inclusive, when signing the ICF
* has a body weight between 50 and 100 kg and a BMI between 18.5 and 30.0 kg/m2, inclusive

Exclusion Criteria:

* Has any current or past clinically meaningful medical or psychiatric condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs, SAEs and AEs leading to discontinuation | up to 16 weeks
  AE: adverse event, SAE: serious adverse event

SECONDARY OUTCOMES:
Cmax | up to 16 weeks
Total IL-6 serum concentrations | up to 16 weeks
Incidence of ADA against ARGX-109 in serum | up to 16 weeks
  ADA: anti-drug antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences - Montreal - Phase I unit, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No